CLINICAL TRIAL: NCT00404794
Title: A Prospective Randomized Open-label Study to Compare Mycophenolate Mofetil and A Prospective Randomized Open-label Study to Compare Mycophenolate Mofetil and Corticosteroid With Tacrolimus and Corticosteroid as Immunosuppressive Treatment for Lupus Membranous Nephritis
Brief Title: A Study to Compare Mycophenolate Mofetil and Tacrolimus in the Treatment of Membranous Lupus Nephritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW05-205 T/868; HARECCTR0500003
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Lupus Nephritis; Glomerulonephritis, Membranous
Keywords: membranous lupus nephritis
MeSH Terms: conditions — Lupus Nephritis; Glomerulonephritis, Membranous | interventions — Prednisolone; Mycophenolic Acid; Tacrolimus

INTERVENTIONS:
Drug: prednisolone and mycophenolate mofetil
Drug: prednisolone and tacrolimus

SUMMARY:
This is a prospective randomized open-label pilot study to compare mycophenolate mofetil in combination with corticosteroid treatment and tacrolimus in combination with corticosteroid treatment in membranous lupus nephritis. The change in urine protein excretion will be the primary outcome studied. The study duration will be 24 months for each patient.

ELIGIBILITY:
Inclusion Criteria:

* abnormal urine protein excretion and biopsy-proven membranous lupus nephritis

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-11; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Proteinuria

SECONDARY OUTCOMES:
Adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Daniel TM Chan, Prof, Principal Investigator — Department of Medicine, Queen Mary Hospital
Locations (1):
- Queen Mary Hospital, Hong Kong, China